CLINICAL TRIAL: NCT03685318
Title: Effect of Shortening the Palatal Extension of the Mouthguard on the Degree of Satisfaction of Water Polo Players: A Randomized Crossover Study
Brief Title: Effect of Shortening the Palatal Extension of the Mouthguard on the Degree of Satisfaction of Water Polo Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jordi Martinez-Gomis, Associate Professor DDS. PhD, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HOUB2018/004
Record Dates: First submitted 2018-09-10; First posted 2018-09-26 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Mouth Protectors; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional mouthguard (Active Comparator): Use of a conventional custom-made mouthguard while playing water polo for two weeks. The conventional mouthguard is designed with the palatal margin at 6 mm from the cervical line.
  Interventions: Device: Use of conventional mouthguard
- Shortened mouthguard (Active Comparator): Use of a shortened custom-made mouthguard while playing water polo for two weeks. The shortened mouthguard is designed with the palatal margin at 2 mm from the cervical line.
  Interventions: Device: Use of shortened mouthguard

INTERVENTIONS:
Device: Use of conventional mouthguard — Use of a conventional custom-made mouthguard while playing water polo
  Arms: Conventional mouthguard
Device: Use of shortened mouthguard — Use of a shortened custom-made mouthguard while playing water polo
  Arms: Shortened mouthguard

SUMMARY:
This study assessed the influence of a reduction of the palate extension of a custom-made mouthguard on the degree of satisfaction of elite water polo players. Eighteen water polo players wore a custom-made conventional mouthguard or a reduced palate extension mouthguard during the training sessions and for competing for two weeks. The sequence was randomized to obtain one-half of the participants started the first week wearing the conventional mouthguard, and the other half wearing the shortened mouthguard. The participants rated the degree of discomfort in reference to speech, breathing, swallowing, nauseas/vomiting, pressure/pain, loosening, aesthetics, and athletic performance, in a 10-point scale, considering 0 no discomfort and 10 maximum discomfort. After each session, players also rated the perception of protection and the degree of satisfaction in a 10-point scale, considering 0 no protection/satisfaction and 10 maximum protection/satisfaction.

DETAILED DESCRIPTION:
This crossover intervention study aimed to assess the influence of a reduction of the palate extension of a custom-made mouthguard on the degree of satisfaction of elite water polo players. Eighteen water polo players participated in this study. Two different custom-made mouthguards were made, a conventional one and a reduced palate extension mouthguard. They wore them during the training sessions and for competing one type of mouthguard for the first and fourth week and the other type of mouthguard for the second and third week. The sequence was randomized to obtain one-half of the participants started the first week wearing the conventional mouthguard, and the other half wearing the shortened mouthguard. The participants rated the degree of discomfort or inconvenience in reference to speech, breathing, swallowing, nauseas/vomiting, pressure/pain, loosening, aesthetics, and athletic performance, in a 10-point scale, considering 0 no discomfort/inconvenience and 10 maximum discomfort/inconvenience. After each session, players also rated the perception of protection and the degree of satisfaction in a 10-point scale, considering 0 no protection/satisfaction and 10 maximum protection/satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* water polo players playing in maximum Spanish category for the season 2017-2018
* Obtaining written informed consent for participating in the project (model consent form)

Exclusion Criteria:

* Players with dental caries, with periodontitis or with temporomandibular joint pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Degree of satisfaction with the mouthguard | Weeks 1-4
  Participant satisfaction was assessed by asking the question "How satisfied are you with your mouthguard?" using a 0-10 point scale, considering 0= totally dissatisfied and 10= totally satisfied. Players rated the mouthguard just after each training session or after each match.

SECONDARY OUTCOMES:
Degree of interference on speech while using the mouthguard | Weeks 1-4
  The degree of interference on speech while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to speech?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on breathing while using the mouthguard | Weeks 1-4
  The degree of interference on breathing while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to breath?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on swallowing while using the mouthguard | Weeks 1-4
  The degree of interference on swallowing while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes your ability to swallow?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort regarding the gag reflex while using the mouthguard | Weeks 1-4
  The degree of discomfort regarding the gag reflex while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard causes a gag reflex?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort because the mouthguard fits too tight | Weeks 1-4
  The degree of discomfort because the mouthguard fits too tight was assessed by asking the question "How much do you think the mouthguard fits too tight?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of discomfort because the mouthguard fits too loose | Weeks 1-4
  The degree of discomfort because the mouthguard fits too loose was assessed by asking the question "How much do you think the mouthguard fits too loose?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on aesthetics while using the mouthguard | Weeks 1-4
  The degree of interference on aesthetics while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes on aesthetics?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of interference on athletic performance while using the mouthguard | Weeks 1-4
  The degree of interference on athletic performance while using the mouthguard was assessed by asking the question "How much do you think wearing the mouthguard interferes athletic performance?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.
Degree of protection with the mouthguard | Weeks 1-4
  The degree of protection perceived by the participant was assessed by asking the question "How much do you feel protected when you are wearing the mouthguard?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Players rated the mouthguard just after each training session or after each match.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Martinez-Gomis, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zamora-Olave C, Willaert E, Montero-Blesa A, Riera-Punet N, Martinez-Gomis J. Risk of orofacial injuries and mouthguard use in water polo players. Dent Traumatol. 2018 Dec;34(6):406-412. doi: 10.1111/edt.12434. Epub 2018 Oct 10. PMID 30156365
- [Background] Gebauer DP, Williamson RA, Wallman KE, Dawson BT. The effect of mouthguard design on respiratory function in athletes. Clin J Sport Med. 2011 Mar;21(2):95-100. doi: 10.1097/JSM.0b013e31820428b0. PMID 21358498
- [Background] Maeda Y, Machi H, Tsugawa T. Influences of palatal side design and finishing on the wearability and retention of mouthguards. Br J Sports Med. 2006 Dec;40(12):1006-8. doi: 10.1136/bjsm.2006.030874. Epub 2006 Sep 25. PMID 17000712
- [Background] Lloyd JD, Nakamura WS, Maeda Y, Takeda T, Leesungbok R, Lazarchik D, Dorney B, Gonda T, Nakajima K, Yasui T, Iwata Y, Suzuki H, Tsukimura N, Churei H, Kwon KR, Choy MMH, Rock JB. Mouthguards and their use in sports: Report of the 1st International Sports Dentistry Workshop, 2016. Dent Traumatol. 2017 Dec;33(6):421-426. doi: 10.1111/edt.12375. PMID 28965361
- [Background] Parker K, Marlow B, Patel N, Gill DS. A review of mouthguards: effectiveness, types, characteristics and indications for use. Br Dent J. 2017 Apr 21;222(8):629-633. doi: 10.1038/sj.bdj.2017.365. PMID 28428580
- [Result] Gomez-Gimeno A, Zamora-Olave C, Cordobes-Navarro M, Willaert E, Martinez-Gomis J. Satisfaction with shortening the palatal extension of a mouthguard for water polo players: A randomized crossover study. Dent Traumatol. 2019 Apr;35(2):135-141. doi: 10.1111/edt.12455. Epub 2019 Jan 7. PMID 30481393